CLINICAL TRIAL: NCT01484236
Title: National Lymphangioleiomyomatosis Registry, France
Acronym: RE-LAM-CE
Status: Recruiting | Type: Observational
Sponsor: Vincent COTTIN (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor-Investigator, Vincent COTTIN, Professor V. Cottin, Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires
Organization: Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires (Other)
Other Study IDs: GERMOP-003
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Lymphangioleiomyomatosis
Keywords: Lymphangioleiomyomatosis
MeSH Terms: conditions — Lymphangioleiomyomatosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
RE-LAM-CE is a registry of lymphangioleiomyomatosis cases in France. its aim is to determine the incidence and prevalence of lymphangioleiomyomatosis in France, including demographic information and information concerning the timing and modalities of diagnosis.

Based on the registry, we will set up a prospective cohort of patients. The database will include detailed medical information, particularly regarding progression of the respiratory function.

DETAILED DESCRIPTION:
Lymphangioleiomyomatosis is a rare pulmonary disease occuring preferentially in women. Few data are available regarding the epidemiology of this disease, the frequency of the various forms with mild to moderate or severe disease, and the rapid or slow progression.

Several sources of information will be used in order to increase completeness. The registry will also allow to estimate the proportion of patients with lymphangioleiomyomatosis who are managed by the Reference Center and Competence Centers for rare lung diseases in France.

Data will be collected by a research assistant, and the study will be coordinated by the Pole IMER - Department of Public health and Epidemiology of HCL (Lyon Hospitals).

This study will provide a better knowledge on the natural course of the disease and the variability in severity and progression of lymphangioleiomyomatosis, and the applicability of diagnostic criteria proposed in 2009. This study will provide the first detailed epidemiological information on Lymphangioleiomyomatosis, will assess the management of this rare disease within the French National Plan for rare diseases 2005 - 2009, and will provide valuable medical information prior to the establishment of clinical trials

ELIGIBILITY:
Inclusion Criteria:

* Patients with sporadic lymphangioleiomyomatosis or associated with Tuberous sclerosis.
* patients diagnosed or hospitalized or seen in consultation since 01/01/2008

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lymphangioleiomyomatosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of cases | 4 years
  Determine incidence and prevalence of lymphangioleiomyomatosis.

SECONDARY OUTCOMES:
localisation of cases | 4 years
  Estimate the proportion of patients with lymphangioleiomyomatosis who are managed by the Reference Center and Centers of excellence for rare lung diseases in France (coverage rate of centers)
Progression-free survival | 4 years
  Determine the frequency of the various forms with mild to moderate or severe, and rapid or slow evolution.
Progression-free survival | 4 years
  Determine applicability of diagnostic criteria proposed in 2009

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Cottin, MD, Principal Investigator — Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires, HCL
Locations (1):
- Hôpital Louis Pradel, Lyon, France

IPD SHARING:
Plan to Share IPD: No